CLINICAL TRIAL: NCT07287332
Title: BLOOM: Pragmatic Feasibility Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erin Barreto, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-004564
Record Dates: First submitted 2025-11-20; First posted 2025-12-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Sepsis; Infection
Keywords: Beta-lactam antibiotics; Sepsis; Septic shock; Pharmacokinetics; Personalized medicine; Therapeutic drug monitoring; Infectious disease
MeSH Terms: conditions — Sepsis; Infections; Shock, Septic; Communicable Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Up-front individualized dosing algorithm (Experimental): Clinical decision support to encourage use of an individualized cefepime dosing algorithm based on eGFRcr-cysC and weight.
  Interventions: Other: Up-front individualized dosing algorithm
- Usual Care (Active Comparator): The standard of care group will receive empiric dosing of cefepime, using an institutional antimicrobial guide based on four categories of eGFRcr.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Up-front individualized dosing algorithm — An individualized cefepime dosing algorithm will be used to determine the cefepime dose and interval. The dose recommendation will be provided using the EHR-prompts to the clinical care team and ordered and/or verified by the ICU pharmacist using an established collaborative practice agreement. As a pragmatic trial, at any point care teams may modify the empiric or subsequent dose based on their clinical judgement.
  Arms: Up-front individualized dosing algorithm
Other: Usual Care — The standard of care group will receive empiric dosing guided by an institutional antimicrobial guide. Cefepime is typically dosed at 0.5-2 g every 8-24 h according to categorical thresholds of estimated creatinine clearance (eGFRcr). Cystatin C and eGFRcr-cys can be calculated and used at clinicians' discretion to aid in drug dose determination.
  Arms: Usual Care

SUMMARY:
The goal of this study is to compare two different ways of dosing cefepime, an antibiotic for very sick patients - the usual approach to dosing or a new dosing method. The new dosing method uses only doses that are available in normal care, but choosing between the different doses is based on more information about the patient's body including their kidney function. The primary purpose of this study is to test how easy it is for healthcare professionals to use the new dosing method and how best to conduct the trial. The study will also assess if the new dosing method helps patients recover faster and reduces side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Admitted to one of the ICUs at the study center
* Prescribed cefepime therapy by the care team

Exclusion Criteria:

* Individuals will be those with a cephalosporin allergy
* Received >1 dose of cefepime in the 24 hours before ICU admission
* Transferred from an external hospital without compatible EHR
* Does not have a cystatin C and a creatinine available for drug dosing
* Acute kidney injury stage 2 or higher
* Receiving renal replacement therapy
* Treated with extracorporeal membrane oxygenation
* Undergoing molecular adsorbent recirculating therapy at the time of beta-lactam initiation
* Pregnant
* Incarcerated
* Declined Minnesota research authorization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients screened who qualified for the study | 1 year or once the sample size is achieved
  Number of patients who quality for the study out of total number of patients screened, reported as a percentage
Distribution of qualified patients across care teams | 1 year or once the sample size is achieved
  Number of patients from each ICU care team who qualify for the study
Adherence to dosing recommendations | 1 year or once the sample size is achieved
  Total number of patients randomized to the up-front individualized dosing algorithm who are prescribed the algorithm's recommended dosage

SECONDARY OUTCOMES:
Number of antibiotic-free days | 28-days
  Number of antibiotic-free days for the first 28 days
ICU length of stay | 1 year
  Number of days of initial ICU stay
Proportion of patients who experience new anti-Pseudomonal beta-lactam resistance | 6 months
  New anti-Pseudomonal beta-lactam resistance which develops within the 6 months following initial treatment
Proportion of patients who experience clinical success | 8 days
  Complete or partial resolution of clinical signs and symptoms attributed to infection across 8 days of therapy.
Proportion of patients who experience microbiologic success | 8 days
  Presumed or documented eradication of causative microorganisms
Mortality | 28-days
  All cause death

CONTACTS AND LOCATIONS:
Overall Officials: Erin Barreto, PharmD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barreto EF, Scheetz MH, Chang J, Cole KC, Fogelson LA, Paul J, Jannetto PJ, Gajic O, Rule AD; Beta Lactam Optimization and Outcomes Management (BLOOM) Study Group. Cystatin C-Guided Dosing Nomogram Improves Target Attainment for Cefepime in the Critically Ill. Crit Care Med. 2025 Apr 1;53(4):e941-e952. doi: 10.1097/CCM.0000000000006622. Epub 2025 Feb 27. PMID 40013864